CLINICAL TRIAL: NCT06091085
Title: Acetazolamide as a Means to Mitigate Falling Ventilatory Drive and Drive-dependent OSA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Scott Aaron Sands, Assistant Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023P002472
Record Dates: First submitted 2023-10-16; First posted 2023-10-19 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: OSA
MeSH Terms: interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: 4-week open-label acetazolamide extension and optional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Acetazolamide (Experimental): Acetazolamide administered for 3 nights, half-dose (1 pill) on the first night followed by full dose (2x250mg pills) for 2 nights
  Interventions: Drug: Acetazolamide
- Placebo (Placebo Comparator): Placebo sugar pills administered for 3 nights, half-dose (1 pill) on the first night followed by full dose (2 pills) for 2 nights
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetazolamide — Administered for 3 nights, half-dose (1 pill) on the first night followed by full dose (2x250mg pills) for 2 nights
  Arms: Acetazolamide
Drug: Placebo — Placebo sugar pills administered for 3 nights, half-dose (1 pill) on the first night followed by full dose (2 pills) for 2 nights
  Arms: Placebo

SUMMARY:
Obstructive sleep apnea (OSA) is a highly prevalent disorder that has major consequences for cardiovascular health, neurocognitive function, risk of traffic accidents, daytime sleepiness, and quality of life. For years, a "classic" model of OSA has been used to describe the disorder, which fails to capture it's complexity. Recently, a model for OSA called drive-dependent OSA was discovered be more prevalent in the OSA population. This drive-dependent OSA is due to ventilation instability that occurs during respiratory events however these individuals have spontaneous increases in drive during respiratory events that stabilize their airway (i.e., via improving upper airway muscle activity) and reduce the risk of respiratory events in people with OSA. Therefore, by stabilizing the ventilatory drive, OSA should be treatable. Acetazolamide is a pharmacological ventilatory stimulant and has been previously shown to reduce OSA severity. As such in this study, the goal is to demonstrate acetazolamide improves OSA severity in 'drive-dependent' OSA people by improving drive-related pharyngeal obstructions compared to the 'classic' OSA people.

DETAILED DESCRIPTION:
The goal of this detailed randomized controlled mechanistic clinical study, with gold-standard measurements of ventilatory drive and dilator muscle activity, is to test the hypotheses that acetazolamide improves OSA in patients with (N=18) but not without (N=18) drive-dependent OSA (i.e. drive-dependent status explains treatment efficacy). We will also show that acetazolamide efficacy is explained by mitigating drive-related reduction in pharyngeal obstruction. A 4-wk open-label extension will explore repeated-dose efficacy without invasive measurements in both subgroups.

Subjects will attend a virtual Screening and Consent visit to assess eligibility for enrollment. Participants will take part in a video call with the consenting doctor to obtain consent (Zoom).

After consent, subjects will first attend a baseline routine sleep study to confirm eligibility (apnea-hypopnea index >15 events/hr) and establish the baseline characteristics. Patients will subsequently attend a specialized physiology night with additional gold-standard measurement of ventilation, ventilatory drive, genioglossus muscle activity, which will serve to establish drive-dependent status.

Those eligible for the study will receive in randomized order the following:

A) Acetazolamide (2x250mg) B) Placebo

Each agent will be administered for 3 nights (2×250 mg pills or 2 matching placebo pills), with a half dose on night 1 (1 pill, same as our preliminary study). Patients will return to the sleep laboratory on the 3rd night of each period for outcomes data collection. Investigators, physicians, participants and outcomes assessors will be blinded to intervention will be blinded to allocation until study completion.

Studies will be 1 week apart (i.e. 3-day treatment, 4-day washout). Adverse event data will be carefully collated.

An open-label extension period (4-weeks) will examine whether differences in acetazolamide efficacy persist with repeated doses between drive-dependent and classic OSA, in the absence of invasive instrumentation (routine sleep equipment only). A 4-week duration is considered the minimum duration necessary for reliable assessment of short-term repeated-dose efficacy and effects on symptoms (e.g. Epworth Sleepiness scale assesses sleepiness over the last month).

Data Analysis

Apneas, hypopneas, sleep stages and arousals from sleep will be scored using current AASM guidelines (hypopneas defined by at least a 30% reduction in airflow in conjunction with either 3% desaturation or arousal) by a technician blinded to the study condition.

Briefly, breath-by-breath values of ventilation and ventilatory drive during sleep are tabulated for the entire night (arousals excluded). Data are sorted into 10-bins (deciles) of ascending drive, and are plotted graphically to show how ventilation ("Flow", median[IQR]) changes with increasing ventilatory drive ("Drive"). We note that functional collapsibility is represented as the value of Flow at normal Drive (100%eupnea), and functional upper airway muscle effectiveness is represented by the slope of the curve. The arousal threshold is represented as the median value of drive preceding scored arousals. Loop gain, not drawn for focus, is calculated as the reduction in Drive that occurs in response to a prior increase in Flow). Plots will be constructed at Baseline, on Acetazolamide, and Placebo for each patient. These plots provide a means to interpret the physiological mechanisms of action of any intervention.

Statistical Analysis Plan

Efficacy by subgroup. Although the study is a mechanistic trial, an intention-to-treat (ITT) analysis will be performed; results for individuals who started a period of treatment and discontinued will be imputed using multiple-imputation with chained equations ("MICE"). Reasons for dropouts will be carefully documented to discriminate between potential dropouts due to AEs as opposed to discontinuation for reasons that are clearly unrelated to study medication (scheduling, intolerance of study equipment, COVID-19, family emergency); an independent DSMB will facilitate adjudication.

The quantitative primary outcome variable will be the continuous percent change in apnea-hypopnea index (AHI) from baseline; the difference in this outcome variable between intervention and placebo (i.e. placebo-corrected effect) will be evaluated using linear mixed model analysis. The primary comparison will be whether the placebo-corrected reduction in AHI from baseline with acetazolamide is greater in drive-dependent OSA vs. classic OSA subgroups (per intervention × subgroup interaction, fixed effects). Subject will be included as a random effect, and models will adjust for period and sequence effects (AB or BA, i.e. carryover effects); the approach also enables incorporation of incomplete data. P<0.05 will indicate statistical significance. As appropriate, percent change from baseline will be transformed to provide a symmetric (normal) distribution using y=x/(2-x) whereby a halving and doubling of the outcome variable have the same magnitude of effect on the transformed variable; results will be back-transformed for presentation.

In the absence of a significant interaction, a significant and clinically-meaningful main effect of intervention within drive-dependent OSA, but not within classic OSA, will also be interpreted as a sign of a meaningful subgroup effect, noting that an important goal is to provide a subgroup enriched for responders in a future trial.

We will also report the response rate i.e. percentage of patients who had a 50% percent reduction in AHI. Secondary outcomes will also be assessed using the same mixed model approach (percent change in hypoxic burden, arousal index; absolute change for N1%); variables will be transformed if necessary to provide a normal distribution before analysis. Similar analysis will be performed for the open-label extension period (absolute change from baseline will be used for each subjective outcome variable); changes in subjective outcomes are exploratory and will be used to provide power analysis for a future trial.

Mechanistic analysis: A per-protocol analysis is planned on the basis that the goal is to assess the mechanisms of action of the agents when present in the circulation. The primary quantitative outcome variable is the increase in ventilation measured at "Nadir Drive" (i.e. 1st decile = 5th centile of drive). The absolute change in this variable with acetazolamide versus baseline will be calculated, and the above analysis approach will examine whether acetazolamide-induced increases in drive promote a greater increase in ventilation in drive-dependent vs classic OSA (per intervention × subgroup interaction). We will also use the same approach to describe the changes in ventilation at Median Drive. We will also examine whether traits causing OSA changed similarly with treatment within each subgroup (collapsibility, compensation, loop gain, arousal threshold).

Power analysis: Sample size is based on the primary outcome model: 36 patients will provide 80% power to detect a 25% mean increase in acetazolamide efficacy in drive-dependent vs. classic OSA subgroups (e.g. average responses = 50% and 25% reduction from baseline, placebo corrected). Power is based on an estimated uncertainty of SD=18% (using model residuals from preliminary data; and N=5000 simulations). Although power analysis was based on N=18 patients with drive-dependent OSA and N=18 patients with classic OSA, in the case of a study imbalance, we will seek to study at least N=13 individuals from each subgroup (>1:2 ratio), leaving the total sample at 36. N=13 and N=23 patients respectively will provide 80% power to detect a 26.5% mean increase in acetazolamide efficacy in drive-dependent vs. classic OSA subgroups (e.g. average responses = 50% and 23.5% reduction from baseline, placebo corrected). Power to detect significant efficacy within drive-dependent OSA is >99% (%reduction in AHI from baseline with acetazolamide vs. placebo). Power is >90% to detect a greater increase in ventilation (1st decile value during sleep) in drive-dependent OSA vs. non-drive dependent OSA. Analysis of the open-label extension period will quantify whether the change in outcomes with acetazolamide vs. placebo persists within each subgroup; Power for the drive-dependent group is >99%.

ELIGIBILITY:
Inclusion Criteria:

* Ages 21-80 years
* Suspected OSA (snoring, sleepiness, witnessed apneas, other clinical symptoms) or diagnosed OSA (severity not required)
* Untreated; No use of OSA treatments within 2 weeks of the baseline study. No plans to start OSA treatments for the duration of the study protocol

Exclusion Criteria:

* Any unstable medical condition
* Current use of the study medication.
* Use of ventilatory stimulant or depressant medications that may complicated interpretation of results (including opioids, barbiturates, doxapram, almitrine, theophylline, 4-hydroxybutanoic acid).
* Contraindications for acetazolamide, including:
* Allergies to sulfonamides - e.g. acetazolamide, hydrochlorothiazide, furosemide, sulfasalazine, celecoxib, sumatriptan, and zonisamide.
* closed-angle glaucoma
* adrenal insufficiency
* known electrolyte or acid/base imbalance (hyponatremia, hypokalemia, hyperchloremia, metabolic acidosis, acidemia)
* clinically-significant kidney disorders (eGFR<60 ml/min/1.73m2)
* clinically-significant liver disorders
* Use of more than 500 mg/day of Aspirin, due to the potential for an interaction of acetazolamide and very high doses of Aspirin (acetylsalicylic acid, a salicylate drug)
* Adrenocortical insufficiency
* Low sodium or potassium
* hyperchloremic acidosis
* Conditions likely to affect obstructive sleep apnea physiology: neuromuscular disease or other major neurological disorder, heart failure, or any other unstable major medical condition.
* Respiratory disorders other than obstructive sleep apnea:
* central sleep apnea (>75% of respiratory events scored as central)
* chronic hypoventilation/hypoxemia (awake SaO2 < 92% by oximetry) due to chronic obstructive pulmonary disease or other respiratory conditions
* Conditions likely to increase arousability from sleep: insomnia
* Other sleep disorders that may complicate establishment of sleep: periodic limb movements (periodic limb movement arousal index > 10/hr), narcolepsy, or parasomnias
* For intramuscular electrodes and catheter: allergy to lidocaine
* Highly-sensitive gag reflex. Patients with a self-reported 'highly-sensitive gag reflex', including an affirmative response to 'Do you sometimes gag when brushing your teeth?', will not take part in the physiology studies given the placement of an esophageal catheter
* For intramuscular electrodes: use of aspirin or other oral anti-platelets / anti-coagulants
* For oronasal mask: severe claustrophobia
* Pregnancy or nursing

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage reduction of apnea-hypopnea Index (AHI) with active versus placebo therapy in drive-dependent vs classic OSA groups | 1 night
  The primary efficacy outcome measure is the apnea hypopnea index (3% desaturation or arousal), presented as a percent reduction from baseline. Differences in this measure with active versus placebo therapy will be assessed. The primary comparison will be the difference in this measure in drive-dependent versus classic OSA subgroups.

SECONDARY OUTCOMES:
Hypoxic burden, %.min/hr | 1 night
  the respiratory event-associated area under the desaturation curve from pre-event baseline
Arousal index, events/hr | 1 night
  average number of arousals per hour of total sleep time
N1 sleep, %total sleep time | 1 night
  Percentage of stage 1 sleep as a proportion of total sleep time

CONTACTS AND LOCATIONS:
Overall Officials: Dillon Gilbertson, Study Director — Brigham and Women's Hospital and Harvard Medical School; Scott Sands, PhD, Principal Investigator — Brigham and Women's Hospital and Harvard Medical School
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared freely with collaborating scientists at any time and more broadly to other scientists 12 months following all planned publications using the data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Deidentified data will be shared freely with collaborating scientists at any time and more broadly to other scientists 12 months following all planned publications using the data.
Access Criteria: Requests should be made in writing to the lead investigator.